CLINICAL TRIAL: NCT05141110
Title: A Phase 1 Clinical Trial, Open-label, Randomized Study in Healthy Subjects to Evaluate Pharmacokinetic Characteristics and Safety of NVP-1705 and NVP-1705-R in Healthy Subjects
Brief Title: Evaluation of Pharmacokinetic and Safety of NVP-1705 and NVP-1705-R in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-1705_BE
Record Dates: First submitted 2021-11-21; First posted 2021-12-02 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: single-dose, crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVP-1705 (Experimental): Tablet formulation for oral administration, single dose of NVP-1705 at Day 1
  Interventions: Drug: NVP-1705
- NVP-1705-R (Active Comparator): Tablet formulation for oral administration, single dose of NVP-1705-R at Day 1
  Interventions: Drug: NVP-1705-R

INTERVENTIONS:
Drug: NVP-1705 — NVP-1705
  Arms: NVP-1705
Drug: NVP-1705-R — NVP-1705-R
  Arms: NVP-1705-R

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and safety of NVP-1705 and NVP-1705-R.

DETAILED DESCRIPTION:
Evaluate the pharmacokinetics and safety of NVP-1705 compared to NVP-1705-R

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject, 19 years of age or older
* Subjects who signed informed consent
* Body mass index(BMI) of 18 to 30.0 kg/㎡

Exclusion Criteria:

* Subject who has clinically significant medical history
* Inadequate subject for the clinical trial by the investigator's decision
* Subjects participated in another clinical trial within 6 months prior to the first administration of investigational product

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of Area under the plasma drug concentration-time curve(AUCt) | 0 ~ 48 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of Maximum observed plasma concentration(Cmax) | 0 ~ 48 hours
  Pharmacokinetics parameter derived from plasma

SECONDARY OUTCOMES:
Evaluation pf Area under the plasma drug concentration-time curve from time 0 to infinity(AUC∞) | 0 ~ 48 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of AUCt/AUC∞ | 0 ~ 48 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of Time of peak concentration(Tmax) | 0 ~ 48 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of Terminal phase of Half-life(t1/2) | 0 ~ 48 hours
  Pharmacokinetics parameter derived from plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jae Woo Kim, M.D., Ph.D, Principal Investigator — H+ Yangji hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, Nambusunhwan-ro, South Korea

IPD SHARING:
Plan to Share IPD: No